CLINICAL TRIAL: NCT00581971
Title: Radiosensitization With a COX-2 Inhibitor (Celecoxib), With Chemoradiation for Cancer of the Head and Neck
Brief Title: Radiosensitization With Celecoxib and Chemoradiation for Head and Neck Cancer
Acronym: RAD0201
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pharmacia (Industry)
Responsible Party: Principal Investigator, Sharon Spencer, MD,, Professor - Radiation Oncology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F020703003; Link No: 000276825
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-03

CONDITIONS: Cancer
Keywords: Radiosensitization; COX-2 inhibitor; Celecoxib; Head and Neck Cancer; Chemoradiation
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms | interventions — Celecoxib; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Celecoxib+Carboplatin/Paclitaxel+Radiation Therapy (Experimental)
  Interventions: Drug: celecoxib; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: celecoxib — 400mg bid starting 1 week before radiotherapy and taken through radiotherapy.
  Other Names: Celebrex
Drug: Carboplatin — IV, AUC 2.0, weekly for weeks 1 through 7
  Other Names: Paraplatin
Drug: Paclitaxel — IV 30 mg/m2, weekly for weeks 1 through 7
  Other Names: Taxol
Radiation: Radiation Therapy — 70.2Gy, at 1.8Gy qd, Monday through Friday

SUMMARY:
This is a single-institution, open-label, non-randomized phase IB/II trial of celecoxib administered concurrently with carboplatin, paclitaxel, and radiation therapy in patients with locally advanced or recurrent squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
Treatment for this protocol consists of radiotherapy, 70.2Gy, at 1.8Gy qd, Monday through Friday.Celecoxib 400mg bid is taken during radiotherapy, starting 1 week before radiotherapy. Carboplatin IV, AUC 2.0, weekly for weeks 1 through 7,Paclitaxel 45 mg/m2, weekly for weeks 1 through 7, and Celecoxib 400mg bid, continuing after therapy for two years or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary squamous cell carcinoma arising in the oropharynx, oral cavity, hypopharynx, or larynx. Patients with recurrences after primary surgery (with no history of radiotherapy or chemotherapy) are also eligible.
* The patient has stage III or IV disease, T3 or higher, or N2 or higher, nonmetastatic. Recurrent need not satisfy these staging requirements on restating, but patients must be nonmetastatic, and either be unresectable, medically inoperable, or refuse further surgery.
* Performance status < 2 (ECOG scale) with a life expectancy of > 12 months.
* Age > 19 years.
* The patient is medically fit to tolerate a course of definitive radiation therapy.
* The patient has:

  * adequate hepatic function with bilirubin < 1.5 x upper limit of normal (ULN),
  * transaminases (SGOT and SGPT) may be up to 2.5 x ULN if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are < ULN,
  * adequate renal function with serum creatinine < 1.5 mg/dl (or estimated creatinine clearance of > 50 mL/min),
  * normal serum calcium,
  * adequate hematologic function as: defined by an absolute neutrophil count > 1500/ml, hematocrit > 24 %, and platelet count > 100,000/ml. Patients with hematocrit between 24 % and 30 % should undergo transfusion or treatment with epoetin, and may be enrolled.
* The patient may have had a prior malignancy but must be disease-free for 5 years prior to study entry. A history of superficial non-melanoma skin cancer or in situ carcinoma of the cervix less than three years will be allowed.
* The patient must agree to use effective contraception if procreative potential exists, and continue contraception for at least 3 months following completion of the study.
* Patient must be informed of the investigational nature of the study and sign an informed consent form.

Exclusion Criteria:

* The patient has received radiation therapy previously to the head and neck. Previous radiotherapy for skin cancers of the head and neck are permitted if the fields do not overlap.
* The patient has received prior chemotherapy for head and neck cancer.
* The patient is pregnant or lactating.
* Squamous cell carcinoma arising in the nasopharynx, sinuses, salivary glands, or the primary is unknown.
* Non-squamous histologies (such as adenoid cystic or mucoepidermoid)
* Peripheral neuropathy > Grade 2.
* Serious non-malignant disease (e.g. congestive heart failure, uncontrolled atrial fibrillation, active hepatitis, renal failure or renal transplant).
* Scleroderma or active connective disorder (Lupus)
* Allergy to celecoxib, sulfonamides, or other NSAIDS
* Any underlying psychological condition that would prohibit the understanding and rendering of informed consent.
* Major surgery < 3 weeks prior to study entry

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-09; Primary Completion 2007-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Spencer, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Aisner J, Sinibaldi V, Eisenberger M. Carboplatin in the treatment of squamous cell head and neck cancers. Semin Oncol. 1992 Feb;19(1 Suppl 2):60-5. PMID 1411628
- [Background] Altorki NK, Keresztes RS, Port JL, Libby DM, Korst RJ, Flieder DB, Ferrara CA, Yankelevitz DF, Subbaramaiah K, Pasmantier MW, Dannenberg AJ. Celecoxib, a selective cyclo-oxygenase-2 inhibitor, enhances the response to preoperative paclitaxel and carboplatin in early-stage non-small-cell lung cancer. J Clin Oncol. 2003 Jul 15;21(14):2645-50. doi: 10.1200/JCO.2003.07.127. PMID 12860939
- [Background] Bourhis J, Calais G, Eschwege F. [Chemoradiotherapy of carcinomas of the upper aerodigestive tract]. Cancer Radiother. 1998 Dec;2(6):679-88. doi: 10.1016/s1278-3218(99)80008-0. French. PMID 9922773
- [Background] Bourhis J, Eschwege F. Radiotherapy-chemotherapy combinations in head and neck squamous cell carcinoma: overview of randomized trials. Anticancer Res. 1996 Jul-Aug;16(4C):2397-402. No abstract available. PMID 8816841
- [Background] Brizel DM, Albers ME, Fisher SR, Scher RL, Richtsmeier WJ, Hars V, George SL, Huang AT, Prosnitz LR. Hyperfractionated irradiation with or without concurrent chemotherapy for locally advanced head and neck cancer. N Engl J Med. 1998 Jun 18;338(25):1798-804. doi: 10.1056/NEJM199806183382503. PMID 9632446
- [Background] Chan G, Boyle JO, Yang EK, Zhang F, Sacks PG, Shah JP, Edelstein D, Soslow RA, Koki AT, Woerner BM, Masferrer JL, Dannenberg AJ. Cyclooxygenase-2 expression is up-regulated in squamous cell carcinoma of the head and neck. Cancer Res. 1999 Mar 1;59(5):991-4. PMID 10070952
- [Background] Choy H, Devore RF 3rd, Hande KR, Porter LL, Rosenblatt P, Yunus F, Schlabach L, Smith C, Shyr Y, Johnson DH. A phase II study of paclitaxel, carboplatin, and hyperfractionated radiation therapy for locally advanced inoperable non-small-cell lung cancer (a Vanderbilt Cancer Center Affiliate Network Study). Int J Radiat Oncol Biol Phys. 2000 Jul 1;47(4):931-7. doi: 10.1016/s0360-3016(00)00420-x. PMID 10863062
- [Background] Choy H, DeVore RF 3rd, Hande KR, Porter LL, Rosenblatt P, Yunus F, Schlabach L, Smith C, Shyr Y, LaPorte K, Johnson DH. Preliminary analysis of a phase II study of paclitaxel, carboplatin, and hyperfractionated radiation therapy for locally advanced inoperable non-small cell lung cancer. Semin Oncol. 1997 Aug;24(4 Suppl 12):S12-21-S12-26. PMID 9331115
- [Background] Eisbruch A, Lyden T, Bradford CR, Dawson LA, Haxer MJ, Miller AE, Teknos TN, Chepeha DB, Hogikyan ND, Terrell JE, Wolf GT. Objective assessment of swallowing dysfunction and aspiration after radiation concurrent with chemotherapy for head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):23-8. doi: 10.1016/s0360-3016(02)02712-8. PMID 12007937
- [Background] Eisenberger M, Hornedo J, Silva H, Donehower R, Spaulding M, Van Echo D. Carboplatin (NSC-241-240): an active platinum analog for the treatment of squamous-cell carcinoma of the head and neck. J Clin Oncol. 1986 Oct;4(10):1506-9. doi: 10.1200/JCO.1986.4.10.1506. PMID 3531424
- [Background] Eisenberger M, Jacobs M. Simultaneous treatment with single-agent chemotherapy and radiation for locally advanced cancer of the head and neck. Semin Oncol. 1992 Aug;19(4 Suppl 11):41-6. PMID 1509280
- [Background] Forastiere AA. Paclitaxel (Taxol) for the treatment of head and neck cancer. Semin Oncol. 1994 Oct;21(5 Suppl 8):49-52. PMID 7939763
- [Background] Forastiere AA. Taxoids in head and neck cancer: the American approach. Acta Otorhinolaryngol Belg. 1999;53(3):253-7. PMID 10635404
- [Background] Frost AR, Sparks D, Grizzle WE. Methods of antigen recovery vary in their usefulness in unmasking specific antigens in immunohistochemistry. Appl Immunohistochem Mol Morphol. 2000 Sep;8(3):236-43. doi: 10.1097/00129039-200009000-00011. PMID 10981877
- [Background] Fu KK, Pajak TF, Trotti A, Jones CU, Spencer SA, Phillips TL, Garden AS, Ridge JA, Cooper JS, Ang KK. A Radiation Therapy Oncology Group (RTOG) phase III randomized study to compare hyperfractionation and two variants of accelerated fractionation to standard fractionation radiotherapy for head and neck squamous cell carcinomas: first report of RTOG 9003. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):7-16. doi: 10.1016/s0360-3016(00)00663-5. PMID 10924966
- [Background] Gaffney DK, Holden J, Zempolich K, Murphy KJ, Dicker AP, Dodson M. Elevated COX-2 expression in cervical carcinoma: reduced cause-specific survival and pelvic control. Am J Clin Oncol. 2001 Oct;24(5):443-6. doi: 10.1097/00000421-200110000-00006. PMID 11586093
- [Background] Gately S. The contributions of cyclooxygenase-2 to tumor angiogenesis. Cancer Metastasis Rev. 2000;19(1-2):19-27. doi: 10.1023/a:1026575610124. PMID 11191059
- [Background] Grizzle, W. E., R. B. Myers, et al. (1998). Immunohistochemical evaluation of biomarkers in prostatic and colorectal neoplasia. John Walker's Methods in Molecular Medicine - Tumor Marker Protocols. M. Hanausek and Z. Walaszek. Totowa, NJ, Humana Press, Inc.: 143-160
- [Background] Grizzle, W. E., R. B. Myers, et al. (1998). Factors affecting immunohistochemical evaluation of biomarker expression in neoplasia. John Walker's Methods in Molecular Medicine - Tumor Marker Protocols. M. Hanausek and Z. Walaszek. Totowa, NJ, Humana Press, Inc.: 161-180.
- [Background] Gupta S, Srivastava M, Ahmad N, Bostwick DG, Mukhtar H. Over-expression of cyclooxygenase-2 in human prostate adenocarcinoma. Prostate. 2000 Jan;42(1):73-8. doi: 10.1002/(sici)1097-0045(20000101)42:13.0.co;2-g. PMID 10579801
- [Background] Hanson WR, Houseman KA, Collins PW. Radiation protection in vivo by prostaglandins and related compounds of the arachidonic acid cascade. Pharmacol Ther. 1988;39(1-3):347-56. doi: 10.1016/0163-7258(88)90082-4. No abstract available. PMID 2849133
- [Background] Hanson WR, Thomas C. 16, 16-dimethyl prostaglandin E2 increases survival of murine intestinal stem cells when given before photon radiation. Radiat Res. 1983 Nov;96(2):393-8. PMID 6647767
- [Background] Hida T, Kozaki K, Muramatsu H, Masuda A, Shimizu S, Mitsudomi T, Sugiura T, Ogawa M, Takahashi T. Cyclooxygenase-2 inhibitor induces apoptosis and enhances cytotoxicity of various anticancer agents in non-small cell lung cancer cell lines. Clin Cancer Res. 2000 May;6(5):2006-11. PMID 10815926
- [Background] Horiot JC, Le Fur R, N'Guyen T, Chenal C, Schraub S, Alfonsi S, Gardani G, Van Den Bogaert W, Danczak S, Bolla M, et al. Hyperfractionation versus conventional fractionation in oropharyngeal carcinoma: final analysis of a randomized trial of the EORTC cooperative group of radiotherapy. Radiother Oncol. 1992 Dec;25(4):231-41. doi: 10.1016/0167-8140(92)90242-m. PMID 1480768
- [Background] Houchen CW, Stenson WF, Cohn SM. Disruption of cyclooxygenase-1 gene results in an impaired response to radiation injury. Am J Physiol Gastrointest Liver Physiol. 2000 Nov;279(5):G858-65. doi: 10.1152/ajpgi.2000.279.5.G858. PMID 11052981
- [Background] Hsu AL, Ching TT, Wang DS, Song X, Rangnekar VM, Chen CS. The cyclooxygenase-2 inhibitor celecoxib induces apoptosis by blocking Akt activation in human prostate cancer cells independently of Bcl-2. J Biol Chem. 2000 Apr 14;275(15):11397-403. doi: 10.1074/jbc.275.15.11397. PMID 10753955
- [Background] Jeremic B, Shibamoto Y, Milicic B, Nikolic N, Dagovic A, Aleksandrovic J, Vaskovic Z, Tadic L. Hyperfractionated radiation therapy with or without concurrent low-dose daily cisplatin in locally advanced squamous cell carcinoma of the head and neck: a prospective randomized trial. J Clin Oncol. 2000 Apr;18(7):1458-64. doi: 10.1200/JCO.2000.18.7.1458. PMID 10735893
- [Background] Kawamori T, Rao CV, Seibert K, Reddy BS. Chemopreventive activity of celecoxib, a specific cyclooxygenase-2 inhibitor, against colon carcinogenesis. Cancer Res. 1998 Feb 1;58(3):409-12. PMID 9458081
- [Background] Kishi K, Petersen S, Petersen C, Hunter N, Mason K, Masferrer JL, Tofilon PJ, Milas L. Preferential enhancement of tumor radioresponse by a cyclooxygenase-2 inhibitor. Cancer Res. 2000 Mar 1;60(5):1326-31. PMID 10728694
- [Background] Kokawa A, Kondo H, Gotoda T, Ono H, Saito D, Nakadaira S, Kosuge T, Yoshida S. Increased expression of cyclooxygenase-2 in human pancreatic neoplasms and potential for chemoprevention by cyclooxygenase inhibitors. Cancer. 2001 Jan 15;91(2):333-8. doi: 10.1002/1097-0142(20010115)91:23.0.co;2-n. PMID 11180079
- [Background] Masferrer JL, Leahy KM, Koki AT, Zweifel BS, Settle SL, Woerner BM, Edwards DA, Flickinger AG, Moore RJ, Seibert K. Antiangiogenic and antitumor activities of cyclooxygenase-2 inhibitors. Cancer Res. 2000 Mar 1;60(5):1306-11. PMID 10728691
- [Background] Munro AJ. An overview of randomised controlled trials of adjuvant chemotherapy in head and neck cancer. Br J Cancer. 1995 Jan;71(1):83-91. doi: 10.1038/bjc.1995.17. PMID 7819055
- [Background] Nishimura G, Yanoma S, Mizuno H, Kawakami K, Tsukuda M. A selective cyclooxygenase-2 inhibitor suppresses tumor growth in nude mouse xenografted with human head and neck squamous carcinoma cells. Jpn J Cancer Res. 1999 Oct;90(10):1152-62. doi: 10.1111/j.1349-7006.1999.tb00690.x. PMID 10595745
- [Background] Oshima M, Dinchuk JE, Kargman SL, Oshima H, Hancock B, Kwong E, Trzaskos JM, Evans JF, Taketo MM. Suppression of intestinal polyposis in Apc delta716 knockout mice by inhibition of cyclooxygenase 2 (COX-2). Cell. 1996 Nov 29;87(5):803-9. doi: 10.1016/s0092-8674(00)81988-1. PMID 8945508
- [Background] Pentland AP, Schoggins JW, Scott GA, Khan KN, Han R. Reduction of UV-induced skin tumors in hairless mice by selective COX-2 inhibition. Carcinogenesis. 1999 Oct;20(10):1939-44. doi: 10.1093/carcin/20.10.1939. PMID 10506108
- [Background] Petersen C, Petersen S, Milas L, Lang FF, Tofilon PJ. Enhancement of intrinsic tumor cell radiosensitivity induced by a selective cyclooxygenase-2 inhibitor. Clin Cancer Res. 2000 Jun;6(6):2513-20. PMID 10873107
- [Background] Peterson HI. Tumor angiogenesis inhibition by prostaglandin synthetase inhibitors. Anticancer Res. 1986 Mar-Apr;6(2):251-3. PMID 2423014
- [Background] Pignon JP, Bourhis J, Domenge C, Designe L. Chemotherapy added to locoregional treatment for head and neck squamous-cell carcinoma: three meta-analyses of updated individual data. MACH-NC Collaborative Group. Meta-Analysis of Chemotherapy on Head and Neck Cancer. Lancet. 2000 Mar 18;355(9208):949-55. PMID 10768432
- [Background] Pillsbury HC 3rd, Webster WP, Rosenman J. Prostaglandin inhibitor and radiotherapy in advanced head and neck cancers. Arch Otolaryngol Head Neck Surg. 1986 May;112(5):552-3. doi: 10.1001/archotol.1986.03780050076013. PMID 3513801
- [Background] Pinto LH, Canary PC, Araujo CM, Bacelar SC, Souhami L. Prospective randomized trial comparing hyperfractionated versus conventional radiotherapy in stages III and IV oropharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 1991 Aug;21(3):557-62. doi: 10.1016/0360-3016(91)90670-y. PMID 1869454
- [Background] Reddy BS, Rao CV, Seibert K. Evaluation of cyclooxygenase-2 inhibitor for potential chemopreventive properties in colon carcinogenesis. Cancer Res. 1996 Oct 15;56(20):4566-9. PMID 8840961
- [Background] Rosenthal DI, Carbone DP. Taxol plus radiation for head and neck cancer. J Infus Chemother. 1995 Spring;5(2):46-54. PMID 8521234
- [Background] Ryu HS, Chang KH, Yang HW, Kim MS, Kwon HC, Oh KS. High cyclooxygenase-2 expression in stage IB cervical cancer with lymph node metastasis or parametrial invasion. Gynecol Oncol. 2000 Mar;76(3):320-5. doi: 10.1006/gyno.1999.5690. PMID 10684704
- [Background] Sanchiz F, Milla A, Torner J, Bonet F, Artola N, Carreno L, Moya LM, Riera D, Ripol S, Cirera L. Single fraction per day versus two fractions per day versus radiochemotherapy in the treatment of head and neck cancer. Int J Radiat Oncol Biol Phys. 1990 Dec;19(6):1347-50. doi: 10.1016/0360-3016(90)90342-h. PMID 2262356
- [Background] Sawaoka H, Tsuji S, Tsujii M, Gunawan ES, Sasaki Y, Kawano S, Hori M. Cyclooxygenase inhibitors suppress angiogenesis and reduce tumor growth in vivo. Lab Invest. 1999 Dec;79(12):1469-77. PMID 10616198
- [Background] Schatz, S. P., L. B. Harrison, et al. (1997). Tumors of the nasal cavity and paranasal sinuses, nasopharynx, oral cavity, and oropharynx. Cancer: 741-801.
- [Background] Sheng H, Shao J, Morrow JD, Beauchamp RD, DuBois RN. Modulation of apoptosis and Bcl-2 expression by prostaglandin E2 in human colon cancer cells. Cancer Res. 1998 Jan 15;58(2):362-6. PMID 9443418
- [Background] Socinski MA, Marks LB, Garst J, Sibley GS, Blackstock W, Turrisi A, Herndon J, Zhou S, Anscher M, Crawford J, Shafman T, Rosenman J. Carboplatin/paclitaxel or carboplatin/vinorelbine followed by accelerated hyperfractionated conformal radiation therapy: a preliminary report of a phase I dose escalation trial from the Carolina Conformal Therapy Consortium. Oncologist. 2001;6 Suppl 1:20-4. doi: 10.1634/theoncologist.6-suppl_1-20. PMID 11182001
- [Background] Soslow RA, Dannenberg AJ, Rush D, Woerner BM, Khan KN, Masferrer J, Koki AT. COX-2 is expressed in human pulmonary, colonic, and mammary tumors. Cancer. 2000 Dec 15;89(12):2637-45. doi: 10.1002/1097-0142(20001215)89:123.0.co;2-b. PMID 11135226
- [Background] Staar S, Rudat V, Stuetzer H, Dietz A, Volling P, Schroeder M, Flentje M, Eckel HE, Mueller RP. Intensified hyperfractionated accelerated radiotherapy limits the additional benefit of simultaneous chemotherapy--results of a multicentric randomized German trial in advanced head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1161-71. doi: 10.1016/s0360-3016(01)01544-9. PMID 11483325
- [Background] Steinauer KK, Gibbs I, Ning S, French JN, Armstrong J, Knox SJ. Radiation induces upregulation of cyclooxygenase-2 (COX-2) protein in PC-3 cells. Int J Radiat Oncol Biol Phys. 2000 Sep 1;48(2):325-8. doi: 10.1016/s0360-3016(00)00671-4. PMID 10974444
- [Background] Steinbach G, Lynch PM, Phillips RK, Wallace MH, Hawk E, Gordon GB, Wakabayashi N, Saunders B, Shen Y, Fujimura T, Su LK, Levin B, Godio L, Patterson S, Rodriguez-Bigas MA, Jester SL, King KL, Schumacher M, Abbruzzese J, DuBois RN, Hittelman WN, Zimmerman S, Sherman JW, Kelloff G. The effect of celecoxib, a cyclooxygenase-2 inhibitor, in familial adenomatous polyposis. N Engl J Med. 2000 Jun 29;342(26):1946-52. doi: 10.1056/NEJM200006293422603. PMID 10874062
- [Background] Suntharalingam M, Haas ML, Conley BA, Egorin MJ, Levy S, Sivasailam S, Herman JM, Jacobs MC, Gray WC, Ord RA, Aisner JA, Van Echo DA. The use of carboplatin and paclitaxel with daily radiotherapy in patients with locally advanced squamous cell carcinomas of the head and neck. Int J Radiat Oncol Biol Phys. 2000 Apr 1;47(1):49-56. doi: 10.1016/s0360-3016(00)00408-9. PMID 10758304
- [Background] Suntharalingam M, Haas ML, Van Echo DA, Haddad R, Jacobs MC, Levy S, Gray WC, Ord RA, Conley BA. Predictors of response and survival after concurrent chemotherapy and radiation for locally advanced squamous cell carcinomas of the head and neck. Cancer. 2001 Feb 1;91(3):548-54. doi: 10.1002/1097-0142(20010201)91:33.0.co;2-a. PMID 11169937
- [Background] Sunwoo JB, Herscher LL, Kroog GS, Thomas GR, Ondrey FG, Duffey DC, Solomon BI, Boss C, Albert PS, McCullugh L, Rudy S, Muir C, Zhai S, Figg WD, Cook JA, Mitchell JB, Van Waes C. Concurrent paclitaxel and radiation in the treatment of locally advanced head and neck cancer. J Clin Oncol. 2001 Feb 1;19(3):800-11. doi: 10.1200/JCO.2001.19.3.800. PMID 11157034
- [Background] Tsujii M, Kawano S, DuBois RN. Cyclooxygenase-2 expression in human colon cancer cells increases metastatic potential. Proc Natl Acad Sci U S A. 1997 Apr 1;94(7):3336-40. doi: 10.1073/pnas.94.7.3336. PMID 9096394
- [Background] Tucker ON, Dannenberg AJ, Yang EK, Zhang F, Teng L, Daly JM, Soslow RA, Masferrer JL, Woerner BM, Koki AT, Fahey TJ 3rd. Cyclooxygenase-2 expression is up-regulated in human pancreatic cancer. Cancer Res. 1999 Mar 1;59(5):987-90. PMID 10070951
- [Background] Vokes EE, Weichselbaum RR, Mick R, McEvilly JM, Haraf DJ, Panje WR. Favorable long-term survival following induction chemotherapy with cisplatin, fluorouracil, and leucovorin and concomitant chemoradiotherapy for locally advanced head and neck cancer. J Natl Cancer Inst. 1992 Jun 3;84(11):877-82. doi: 10.1093/jnci/84.11.877. PMID 1375657
- [Background] Yoshimura R, Sano H, Masuda C, Kawamura M, Tsubouchi Y, Chargui J, Yoshimura N, Hla T, Wada S. Expression of cyclooxygenase-2 in prostate carcinoma. Cancer. 2000 Aug 1;89(3):589-96. PMID 10931458

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib + Carboplatin/Paclitaxel+Radiation Therapy: Patients with locally advanced head and neck cancer will be treated with weekly carboplatin, paclitaxel, and concurrent radiotherapy. Radiotherapy will be delivered at 1.8 Gy every day, to a maximum dose of 70.2 Gy. Carboplatin will be dosed at AUC=2.0, while paclitaxel will be dosed at 30mg/m2. Celecoxib will be delivered at 400mg twice daily, starting 1 week prior to the onset of radiotherapy to establish constant blood levels.
Period: Overall Study
Arm/Group | Celecoxib + Carboplatin/Paclitaxel+Radiation Therapy
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Celecoxib + Carboplatin/Paclitaxel+Radiation Therapy
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 53.83 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Toxicity of Celecoxib With Concurrent Weekly Chemotherapy and Radiotherapy in the Treatment of Locally Advanced or Recurrent Squamous Cell Carcinoma of the Head and Neck.
Description: Particpants experiencing Acute Toxicities > Grade 3
Time Frame: 2 years from radiation therapy
Measure: Number; unit: participants
Groups:
- Acute Toxicity: Participants that experienced Grade 3 or higher toxicity factors.
Arm/Group | Acute Toxicity
Number analyzed (Participants) | 30
participants
  Hematologic | 12
  Dermatitis | 7
  Mucositis/Dysphagia | 16

2. Primary Outcome: Response as Evaluated by Recurrence of Diseases
Description: Evaluate the response to concurrent celecoxib, carboplatin, paclitaxel, and radiotherapy in the treatment of locally advanced SSC of the head and neck. Response is determined by local control only, local and distant metastasis, distant metastasis only, second primary, and surgical salvage.
Time Frame: 2 years from end of treatment (Radiation therapy)
Measure: Number; unit: Participants
Arm/Group | Recurrence
Number analyzed (Participants) | 14
Participants
  Local Control Only | 6
  Local Control and Distant Metastasis | 2
  Distant Metastatsis Only | 1
  Secondary Primary - Site Unknown | 2
  Surgical Salvage | 3

ADVERSE EVENTS:
Arm/Group | Celecoxib + Carboplatin/Paclitaxel+Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib + Carboplatin/Paclitaxel+Radiation Therapy (N=30)
Stroke (Vascular disorders) | 1 (1)
Febrile Neutropenia (Immune system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (in absence of Neutropenia) (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib + Carboplatin/Paclitaxel+Radiation Therapy (N=30)
Mucositis (Gastrointestinal disorders) | 8 (9)
Neutropenia (Blood and lymphatic system disorders) | 10 (12)
Radiation Dermatitis (Skin and subcutaneous tissue disorders) | 5 (7)
Dysphagia (Gastrointestinal disorders) | 21 (24)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No